CLINICAL TRIAL: NCT06527573
Title: Targeting Anterior or Posterior, Where is Better for DOC
Brief Title: Effects of rTMS With Different Stimulation Spots in Patients With Disorders of Consciousness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Qiuyou Xie, principal investigator, Zhujiang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: L20240725
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Disorder of Consciousness
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active repetitive transcranial magnetic stimulation on prefrontal lobes (Experimental): Real stimulation will be delivered on individualized target using a real coil
  Interventions: Device: active repetitive transcranial magnetic stimulation
- Active repetitive transcranial magnetic stimulation on posterior parietal lobes (Experimental): Real stimulation will be delivered on individualized target using a real coil
  Interventions: Device: active repetitive transcranial magnetic stimulation
- Sham repetitive transcranial magnetic stimulation (Sham Comparator): Sham stimulation will be delivered on individualized target using a sham coil
  Interventions: Device: sham repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: active repetitive transcranial magnetic stimulation — During the rTMS-active stage, treatment will be given for 7 consecutive days (two session daily). The participants will be placed in the semi-reclining position on either a normal chair or a wheelchair and each stimulation session will last 20 minutes with a frequency of 10 Hz (train duration: 1s; inter-train interval: 5s; 200 effective stimulation series; 2000 pulses at 90% of RMT).
  Arms: Active repetitive transcranial magnetic stimulation on posterior parietal lobes; Active repetitive transcranial magnetic stimulation on prefrontal lobes
Device: sham repetitive transcranial magnetic stimulation — The sham coil will be used which has no magnetic field to send to the cerebral cortex while appearing to be the same shape as the active coil, with good approximation of auditory feedback.(train duration: 1s; inter-train interval: 5s; 200 effective stimulation series; 0 pulses at 90% of RMT).
  Arms: Sham repetitive transcranial magnetic stimulation

SUMMARY:
Disorders of consciousness are a state in which consciousness is affected by brain damage, resulting in dysfunctions in alertness, awareness, and behavior. Patients with disorders of consciousness can be categorized into coma, unresponsive arousal syndrome（UWS）, and minimally conscious states（MCS）. Common causes include craniocerebral trauma and non-craniocerebral trauma causes such as stroke and ischemic-hypoxic encephalopathy. The number of patients with disorders of consciousness is rapidly increasing worldwide and is not only affecting the lives of individuals and their families, but is becoming a serious public health threat.Transcranial magnetic stimulation uses an electromagnetic pulse to induce focalised neural depolarisation and firing. Repeated transcranial magnetic stimulation, compared with single pulse transcranial magnetic stimulation, can influence brain plasticity and cortical organisation through alterations of neuronal excitability and is now being used to improve consciousness and functional recovery in patients with disorders of consciousness. However, the optimization of TMS stimulation parameters has become one of the key factors affecting the therapeutic efficacy, especially the choice of treatment location.

Method:This study is a randomized double-blind controlled trial.And eighty-four patients are expected to be recruited and they will be randomly assigned in a 1:1:1 ratio to two test groups and one control group of 28 patients each.. Each patient receives a one-week period of repetitive transcranial magnetic stimulation at 10 Hz twice daily for a total of 14 treatments. Primary and secondary evaluation indices will be performed at each baseline and after rTMS treatment. Primary and secondary evaluating indicators will be performed at each baseline and after rTMS treatment. Primary outcome will be determined as behavioral response to treatment as measured using the Coma Recovery Scale - Revised (CRS-R). Resting-state high-density EEG and TMS-EEG will be also recorded to investigate the neurophysiological correlates by rTMS.

Discussion:This study will contribute to the selection of therapeutic target locations for rTMS in patients with disorders of consciousness and has the potential to explore mechanisms of consciousness and to validate the role of rTMS parameter optimization in patients with disorders of consciousness using randomized controlled trials

ELIGIBILITY:
Inclusion Criteria:

1. acquired brain injuries less than 1 year and more than 28 days in DOC;
2. clinical diagnosis of DOC Disease;
3. no medical history of neuropsychiatric diseases;
4. no contraindications for rTMS or EEG, no sedatives in use or other drugs that might interfere with brain stimulation, such as Na+ or Ca2+ channel blockers or NMDA receptor antagonists;
5. stable state of disease and vital signs;
6. the integrity of the individualized stimulation target cortex are verified by MRI.

Exclusion Criteria:

1. patients in other non-invasive or invasive neuroregulation trials;
2. motor evoked potential (MEP) in M1 region cannot be induced by TMS pulse;
3. uncontrolled epilepsy, seizure within 4 weeks before enrollment;
4. metallic implant in the skull, pacemaker, craniotomy under the stimulated site, implanted brain device.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-07-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline JFK Coma Recovery Scale-Revised(CRS-R) | immediately after 7 days rTMS session
  The CRS-R includes six items addressing auditory, visual, motor, oromotor, communication, and arousal processes, each with different response categories, and its total score is calculated considering the presence or absence of specific behavioral responses to sensory stimuli, with a range between 0 (worst) and 23 (best). Each item of CRS-R is in good agreement with the diagnostic and differential diagnostic criteria of VS/UWS, MCS and EMCS. The higher scores mean a better outcome.Secondary outcome

SECONDARY OUTCOMES:
Change from Baseline Resting-State EEG | immediately after 7 days rTMS session
  Based on the assumption that specific cortical oscillations indicate varying levels of thalamocortical integrity that has defined four dynamic regimes that build on the mesocircuit model, each detectable with EEG and corresponding to a thalamo cortical state that indicates progressive circuit recovery.These EEG types are labeled A-D (hence, ABCD model) .Later types (C, D) denote more progressive recovery (i.e., are "better") than earlier types, (A, B), which correspond to a quiescent thalamic state.
Change from Baseline TMS-EEG | immediately after 7 days rTMS session
  Transcranial magnetic stimulation combined with electroencephalography (TMS-EEG) is an effective way to measure cortical activity..In this study, PCIst, a derivative version of PCI, PCIst was chosen as an alternative, which estimates the complexity of TMS perturbations by signal decomposition and recurrence quantification analysis (RQA)

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No